CLINICAL TRIAL: NCT06543381
Title: Pilot Trial of Olutasidenib Maintenance Post Allogeneic Hematopoietic Cell Transplantation in Patients Carrying IDH1 Mutation With AML, MDS, or CMML Disease
Brief Title: Olutasidenib for the Treatment of Patients With IDH1 Mutated AML, MDS or CMML After Donor Hematopoietic Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23483; NCI-2024-06471 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23483 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Specimen Handling; olutasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olutasidenib) (Experimental): Starting 50-120 days after transplant, patients receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Olutasidenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Olutasidenib — Given PO
  Other Names: FT 2102; FT-2102; FT2102; IDH1-R132 Inhibitor FT-2102; Rezlidhia

SUMMARY:
This phase I trial tests the safety, side effects, and effectiveness of olutasidenib in preventing the return of disease (relapse) in patients who have undergone donor (allogeneic) hematopoietic cell transplant for acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myelomonocytic leukemia (CMML) carrying an IDH1 mutation. Olutasidenib is in a class of medications called IDH1 inhibitors. It works by slowing or stopping the growth of cancer cells. Giving olutasidenib may be safe, tolerable and/or effective in preventing relapse in patients with IDH1 mutated AML, MDS or CMML after an allogeneic hematopoietic cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and tolerability of olutasidenib as maintenance therapy after allogeneic hematopoietic cell transplantation (HCT) in patients with IDH1-mutated acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), or chronic myelomonocytic leukemia (CMML).

SECONDARY OBJECTIVES:

I. Assess overall survival (OS) and leukemia-free survival (LFS) at 1 and 2 years after first dose of olutasidenib.

II. Estimate cumulative incidence of relapse (CIR), non-relapse mortality (NRM), graft-versus-host disease (GVHD) free, relapse-free survival (GRFS) at 1 and 2 years after first dose of olutasidenib.

III. Rate and grading of acute GVHD of grades 2-4 and 3-4 at day 100 post allogeneic HCT.

IV. Incidence and grading of chronic GVHD of all grades at 1 and 2 years after first dose of olutasidenib.

EXPLORATORY OBJECTIVES:

I. Monitor disease status by multiparameter flow cytometry among a subset of patients with minimal residual disease (MRD)+ disease when starting olutasidenib.

II. Molecular monitoring of disease status by HopeSeq complete (at City of Hope [COH]) and equivalent next generation sequencing (NGS) assay at Cleveland Clinic.

III. Monitor immune reconstitution by flow cytometry during protocol therapy. IV. Mutant (m)IDH1 testing on peripheral blood samples with standard polymerase chain reaction (PCR).

V. Investigate IFN-ɣ signaling in immune cell subsets before and during maintenance therapy.

VI. Monitor mIDH1 variant allele fraction (VAF) by droplet digital PCR (ddPCR) beads, emulsion, amplification, magnetics (BEAM)ing technology on peripheral blood.

OUTLINE:

Starting 50-120 days after bone marrow transplant, patients receive olutasidenib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days and then up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies. If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2 or Karnofsky performance status (KPS) ≥ 70
* Patients who are scheduled to receive or have already undergone allogeneic hematopoietic cell transplantation (alloHCT) from any donor type, any conditioning regimen, and regardless of GVHD prophylaxis will be include
* Patients must have AML, MDS, or CMML with mIDH1 diagnosis at diagnosis (regardless of time from HCT). Note: Patient with pre-HCT disease relapse will no be included if mIDH1 is not detected after relapse
* Day 30 marrow post alloHCT should show evidence of morphologic remission with < 5% bone marrow (BM) blasts. Patients with MRD-positive status either by flow cytometry or IDH1 mutation testing will be eligible
* Patients with previous therapy with IDH1 inhibitors will be included
* Absolute neutrophil count (ANC) > 1000/mm^3 (within 28 days prior to day 1 of protocol)
* Hemoglobin ≥ 8.0 gm/dL (within 28 days prior to day 1 of protocol)
* Platelets ≥ 50,000/mm^3 (within 28 days prior to day 1 of protocol) Note: Patients with lower counts can enroll if infection cytomegalovirus (CMV)/human herpes virus 6 (HHV6), etc. is being treated actively
* Bilirubin ≤ 2 x upper limit of normal (ULN) (within 28 days prior to day 1 of protocol) (unless has Gilbert's disease). Patients with abnormal liver function tests (LFTs) due to active GVHD will not be eligible
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2 x ULN (within 28 days prior to day 1 of protocol). Patients with abnormal LFTs due to active GVHD will not be eligible
* Creatinine clearance of ≥ 30/min/1.73 m^2 for participants with creatinine levels above institutional normal per 24 hour urine test or the Cockcroft-Gault formula (within 28 days prior to day 1 of protocol)
* Corrected QT interval (QTc) ≤ 480 ms (Note: To be performed within 28 days prior to day 1 of protocol therapy)
* Seronegative for HIV antigen/antibody (Ag/Ab) combo, hepatitis C virus (HCV) (if positive, hepatitis C ribonucleic acid [RNA] quantitation must be performed), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (within 28 days prior to day 1 of protocol)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 28 days prior to day 1 of protocol). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential, defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only), to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

Exclusion Criteria:

* Patients with more than one allogeneic HCT
* History of allergic reactions attributed to compounds of similar chemical or biological composition to study agent
* Active diarrhea considered clinically significant and may impair oral drug administration
* Clinically significant uncontrolled illness
* Uncontrolled infection requiring systemic antimicrobials

  * Active infection: Patients with treated viral, bacterial or fungal infections that are controlled on therapy will be allowed to participate
* Participant has detectable human immunodeficiency virus (HIV) viral load within the previous 6 months (must have viral load testing prior to study enrollment if participant has a known history of HIV 1/2 antibodies)
* Active hepatitis B or C, or HIV
* Other active malignancy. Participants with history of prior malignancy treated with curative intent who achieved CR more than 2 years before study entry are eligible. This exclusion rule does not apply to non-melanoma skin tumors and in-situ cervical cancer
* Females only: Pregnant or breastfeeding
* Active grade II-IV acute GVHD per Mount Sinai Acute Graft Versus Host Disease International Consortium (MAGIC) criteria and/or requiring systemic steroids with prednisone dose equivalent of ≥ 0.25 mg/kg at end of 4 weeks. Patients with a mild form of acute GVHD involving skin, gut or liver requiring topical steroid creams or oral beclomethasone (8 mg/day), entocort, (9 mg/day) and/or solumedrol (and equivalent prednisone) will be allowed
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Proportion of patients completing at least 6 months of study therapy | Up to 2 years
  Tolerability will be defined as the proportion of patients who complete at least 6 months of study therapy.

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment to death, assessed up to 2 years
  OS will be analyzed using the Kaplan-Meier method.
Leukemia-free survival (LFS) | From start of treatment to relapse or death, assessed up to 2 years
  LFS will be analyzed using the Kaplan-Meier method.
Time to relapse | From start of treatment to relapse, assessed up to 2 years
  Time to relapse will be analyzed using the curves of cumulative incidence.
Non-relapse mortality (NRM) | From start of treatment to death from causes other than relapse, assessed up to 2 years
  NRM will be analyzed using the curves of cumulative incidence.
Graft versus host disease (GVHD) free, relapse-free survival (GRFS) | From start of treatment to grade III or IV acute GVHD, chronic GVHD requiring systemic therapy, relapse, or death, assessed up to 2 years
  GRFS will be analyzed using the Kaplan-Meier method.
Rate of acute GVHD (aGVHD) grades II-IV and III-IV | From transplant to aGVHD onset, assessed up to 2 years
  Rate of aGVHD will be graded according to Mount Sinai Acute Graft Versus Host Disease International Consortium Grading System grading.
Incidence of chronic GVHD (cGVHD) | From start of treatment to cGVHD onset, assessed up to 2 years
  Incidence of cGVHD will be scored according to National Institutes of Health Consensus Staging and will be measured from start of protocol therapy to the documented/biopsy proven cGVHD onset date.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Cleveland Clinic Cancer Center, Cleveland, Ohio